CLINICAL TRIAL: NCT05444413
Title: Effect of Ultrasound-guided Platelet-Rich Plasma Nerve Block Combined With Drugs in the Treatment of Intractable Postherpetic Neuralgia
Brief Title: Platelet-rich Plasma in the Treatment of Intractable Postherpetic Neuralgia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Yuan Zhou, Deputy chief physician, Affiliated Hospital of Nantong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-K036
Record Dates: First submitted 2022-06-23; First posted 2022-07-05 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: PHN - Post-Herpetic Neuritis
Keywords: platelet-rich plasma; Intractable postherpetic neuralgia

STUDY DESIGN:
Intervention Model Description: patients with Intractable Postherpetic Neuralgia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ultrasound-guided platelet rich plasma nerve block combined with drugs (Experimental): selected patients were treated by the ultrasound-guided platelet rich plasma nerve block once a week for the 4 consecutive weeks while they were given the regular medicine which are taking pregabalin and amitriptyline hydrochloride orally, and the dosage shall be increased or decreased according to the patient's condition.
  Interventions: Biological: ultrasound-guided platelet rich plasma nerve block

INTERVENTIONS:
Biological: ultrasound-guided platelet rich plasma nerve block — selected persons are treated by ultrasound-guided platelet rich plasma nerve block and the regular medicine

SUMMARY:
used ultrasound-guided platelet rich plasma nerve block to treat Intractable Postherpetic Neuralgia.

DETAILED DESCRIPTION:
Postherpetic neuralgia (PHN) is a kind of pain caused by varicella zoster virus invading the human body and infecting the corresponding ganglia. The affected ganglia are inflamed or even necrotic, affecting the nerve endings, the dorsal horn of the spinal cord and the sensory nerve tissues below, and the course of the disease is more than one month or more. Most patients can avoid PHN by timely and effective treatment in the acute herpes zoster period. However, some patients with intractable postherpetic neuralgia fail to receive timely and effective pain control treatment in the early stage of the disease, and the current commonly used clinical treatment methods often fail to achieve effective treatment results. Such patients often have a long course of disease, which can last for three to five years or even longer, Nerve damage is also more serious. Long term pain has seriously affected the quality of life of such patients. Therefore, how to quickly and effectively control pain has become the diagnosis and treatment goal of such patients with intractable post herpetic neuralgia. Platelet rich plasma (PRP) was widely used in muscle and bone repair due to its function of promoting tissue repair in the early stage. Recently, it was found that PrP can also promote nerve repair. Therefore, in order to further explore the therapeutic effect of PRP on refractory PHN patients, our department used ultrasound-guided platelet rich plasma nerve block to treat Intractable PHN.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of PHN: have a history of acute herpes zoster, the pain lasts for more than half a year, and there is paroxysmal pain in the affected nerve distribution area;
* Preoperative visual analog scale (VAS) score ≥ 5;
* Those who can cooperate with the treatment;
* We agreed to inject platelet rich plasma into nerve block under the guidance of ultrasound, and signed the informed consent form.

Exclusion Criteria:

* Systemic infection or puncture local infection;
* Serious disturbance of cardiovascular and cerebrovascular function;
* Abnormal bleeding and coagulation function or complicated with blood system diseases;
* Mental disorders;
* Severe dysfunction of important organs in the body

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
The changes from degree of pain that patients feel after the treatment are assessed by the numerical rating scale (NRS). | Change from the numerical rating scale at 6 months
  This method is composed of 11 numbers from 0 to 10. Patients use 11 numbers from 0 to 10 to describe the intensity of pain. (0="no pain"and 10=the "worst pain")

SECONDARY OUTCOMES:
The changes from degree of pain that patients feel after the treatment are also assessed by the Short-form McGill Pain Questionnaire(SF-MPQ). | Change from the total score of Short-form McGill Pain Questionnaire at 6 months
  When evaluating item (1), ask the thinker questions one by one, and mark the corresponding level according to the pain level the thinker answers.
  When evaluating item (2), vas ruler shall be adopted. This ruler is a 10cm long swimming ruler with 10 graduations marked on one side and "0" and "10" at both ends, indicating no pain,"10" represents the most severe pain that the patient can't bear in his life. During clinical use, the side with scale is turned away from the patient, and the patient is asked to mark the corresponding position representing his pain level in the past day on the ruler. The evaluator evaluates the number of patients according to the position marked by the patient (for example, 5.4cm is 5.4 points), and records it in the table.
  When evaluating item (3), mark the corresponding score according to the patient's subjective feelings.
  Finally, the total scores of PRI, vas and PPI were evaluated. （The higher the total score, the more severe the pain）
The changes from degree of the patient' sleep quality after the treatment are assessed by the Athens Insomnia Scale. | Change from the patient' sleep quality at 6 months
  Ask the examinee to carefully review his sleep experience in the past one month for questions ① - ⑧. If it happens to you at least three times a week, circle the corresponding self-assessment results. Then calculate the total score for evaluation.
  Assessment result judgment:
  (1) If the total score is less than 4, there is no sleep disorder: (2) if the total score is 4-6, it is suspected that there is a big sleep; (3) If the total score is above 6: Insomnia

CONTACTS AND LOCATIONS:
Overall Officials: yuan zhou, doctor, Study Director — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No